CLINICAL TRIAL: NCT05249764
Title: Effects of Home-Based Exercise Training on Physical Fitness and Functionality in Sedentary Older Adults During the COVID-19 Pandemic
Brief Title: Home-Based Exercise Training in Older Adults During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Yuruk, PT, PHd, Professor, lecturer in Baskent University, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA2020/116
Record Dates: First submitted 2022-02-17; First posted 2022-02-22 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Physical Inactivity; Aging; COVID-19 Pandemic
Keywords: Exercise; Physical Fitness; Functionality; Older adults
MeSH Terms: conditions — Sedentary Behavior; COVID-19; Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the study and control group do not know the content of the exercise program. All groups are taking exercise programs individually at their home. So that individuals are not aware of the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Exercise program was prepared based on WHO, American College of Sports Medicine (ACSM), Geriatrics Physiotherapists Association and Otago exercise program for the exercise group. The older adults are given individual supervised exercise training in their own homes for eight weeks, 3 days a week and 45 minutes a day, by a physiotherapist according to social distance rules. This exercise training consists of a program that includes strengthening, flexibility, aerobic and balance exercises. Each exercise is started with eight repetitions and each week will be increased by two repetitions. In case of fatigue, a rest is given. Brochures are also be prepared for the exercises. Before each session, individuals performed warm-up exercises for 5 minutes. At the end of the session, individuals performed cooling exercises.
  Interventions: Other: Supervised Home Based Exercise Training
- Control (Active Comparator): Individuals in the control group are performing stretching exercises for proximal extremity muscles for 15 minutes 3 times a week for eight weeks. The participants also perform breathing exercises for 5 minutes a day.
  Interventions: Other: Unsupervised stretching and breathing exercises

INTERVENTIONS:
Other: Supervised Home Based Exercise Training — Exercise program was prepared based on WHO, American College of Sports Medicine (ACSM), Geriatrics Physiotherapists Association and Otago exercise program for the exercise group. The older adults are given individual supervised exercise training in their own homes for eight weeks, 3 days a week and 45 minutes a day, by a physiotherapist according to social distance rules. This exercise training consists of a program that includes strengthening, flexibility, aerobic and balance exercises. Each exercise is started with eight repetitions and each week will be increased by two repetitions. In case of fatigue, a rest is given. Brochures are also be prepared for the exercises. Before each session, individuals performed warm-up exercises for 5 minutes. At the end of the session, individuals performed cooling exercises.
  Arms: Exercise
Other: Unsupervised stretching and breathing exercises — Individuals in the control group are performing stretching exercises for proximal extremity muscles for 15 minutes 3 times a week for eight weeks. The participants also perform breathing exercises for 5 minutes a day.
  Arms: Control

SUMMARY:
The physical fitness and functionality of older adults are affected during the COVID-19 Pandemic. Regular exercise programs are effective in physical fitness and functioning in older adults. Individualized and supervised exercise programs for older adults in a safe environment can improve physical fitness and functionality. This study aims to examine the effect of home-based and exercise training on physical fitness and functionality in sedentary older adults during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Purpose: This study aims to examine the effect of home-based supervised exercise programs on physical fitness and functionality in sedentary older adults during the Covid-19 pandemic.

Methods: The older adults participating in the study are divided into two groups as exercise group and the control group. Individual exercise training is applied to the exercise group for eight weeks, three days a week, and 45 minutes a day. This exercise training consists of a program that includes strengthening, flexibility, aerobic, and balance exercises. The control group is given only of stretching and breathing exercises. Individuals are evaluated using the Berg Balance Scale, Timed Up and Go Test, Senior Fitness Test, and Tinetti Falling Efficacy Scale before starting the study and at the end of the eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged between 65-85 years
2. Individuals have 24 points and above from the Standardized Mini-Mental State Examination
3. Sedentary individuals whose physical activity levels are inactive or minimally active group according to the Short form of International Physical Activity Questionnaire (IPAQ-SF).
4. Individuals who can stand for at least 90 seconds without assistance
5. Individuals who voluntarily agree to participate in the study
6. Individuals who have not suffered from COVID infection.

Exclusion Criteria:

1. Individuals who have malignancy
2. Individuals who are ambulatory with assistance
3. Individuals who have severe vision loss
4. Individuals who have a neurological disease (Stroke, Parkinson, Multiple Sclerosis)
5. Individuals who had surgery in the last six months
6. Individuals who have congestive heart failure
7. Individuals who have received exercise training in the last six months

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline lower extremitu muscle strength at 8 weeks | Before the program and after eight weeks program
  The chair stand test determines the muscle strength of the lower extremities. The older adult seat on a chair without arm support, with his/her feet on the ground and arms cross in the front of the chest. The number of full stands from the seated position perform within 30 seconds is recorded.
Change from baseline upper extremity muscle strength at 8 weeks | Before the program and after eight weeks program
  The arm curl test determines the upper extremity muscle strength. The older adult seat towards the dominant side on a chair without arm support. In this test, older women and men lift weights of 2.27 and 3.63 kilograms, respectively, starting with a full elbow extension with dominant arms and flexing the elbow to full flexion. The total number of lifts perform for 30 seconds is recorded.
Change from baseline aerobic endurance at 8 weeks | Before the program and after eight weeks program
  The 2-minute step test measures the aerobic endurance of the older adults as an alternative to the 6-minute walk test. The distance from the iliac crest to the midpoint of the patella is measured by a tape to determine the knee-stepping height. The midpoint between these two anatomical structures is determined. The height of the determined point from the ground is measured and marked on a wall. The older adult begins stepping as quickly as possible to reach the marked height for two minutes. The total number of correct steps is recorded. If any of the steps (right or left) do not reach the target height, those steps are considered invalid.
Change from baseline lower extremity flexibility at 8 weeks | Before the program and after eight weeks program
  The Chair sit-and-reach test is a modified form of the sit-and-reach test, which determines the flexibility of the hamstring muscle group. The older adult sits on the front of a chair. Then they extend the right or left knee to a full extension, the heel on the floor, and ankle in a neutral position of 90 degrees. The other knee is flexed to approximately 90 degrees. Then, the older adult is asked to reach the toes of the extended limb with his/her same side upper limb. If the middle finger could not reach to the toes, the distance is recorded as a 'minus' score; if it could touch the toes, then a distance of 'zero' score is recorded; and if it could reach past the toes, then the distance is recorded as a 'plus' score.
Change from baseline upper extremity flexibility at 8 weeks | Before the program and after eight weeks program
  The Back scratch test evaluates the flexibility of the upper extremities. The older adult is asked to stand up and place his/her preferred hand over the same shoulder, palm down and fingers extended, and reach down the middle of the back as far as possible. Then the researcher want the older adult to place the other arm around the back of the waist with the palm up and reach up the other hand. The distance between the middle fingers of both hands is measured with a tape. If the middle fingers do not touch each other, the distance is recorded as a 'minus' score, if it reaches the other, then a 'zero' score is recorded as; and if fingers could cross each other, then 'plus' score is recorded.
Change from baseline balance and agility at 8 weeks | Before the program and after eight weeks program
  The 8-foot up and go test determines the dynamic balance and agility of the older adults. The older adult gets up from a chair without any arm support and walk 2.44 meters as quickly as possible; then turn around a cone (at a specified position) and come back to sit down on the chair. The time between the older adults' starting movement and sitting down on the chair is recorded in seconds.

SECONDARY OUTCOMES:
Change from baseline Berg Balance Scale at 8 weeks | Before the program and after eight weeks program
  Berg Balance Scale evaluates the balance and determines fall risk in individuals. The scale assesses 14 tasks involving static and dynamic balance. Each task is given a score ranging from 0 (failed to complete the task) to 4 (performed the task independently). The scores of the 14 tasks are summed to obtain a total score ranging from 0 to 56. 0-20 points indicate balance disorder, 21-40 points indicate acceptable balance skills, 41-56 points indicate good balance.
Change from baseline Timed up and go test at 8 weeks | Before the program and after eight weeks program
  The TUGT includes getting up from a chair, walking, turning, standing and sitting again, and assesses independent mobility and functional ability. Before the test, the individual is asked to get up from the chair, to walk at a safe and normal speed up to the previously marked distance of 3 meters, to turn, to walk backwards, and to sit on the chair. The time elapsed during this time is recorded in seconds.
Change from baseline Tinetti Fall Efficancy Scale at 8 weeks | Before the program and after eight weeks program
  The Tinetti Fall Efficancy Scale assesses effectiveness and safety of individuals while performing daily activities. The scale has 10-items. These items are; going to bed and getting out of bed, sitting and getting out of a chair, bathing, dressing and undressing, lying in the closet, walking around the house, looking at the door or phone, preparing food, tidying the house, and shopping. In the scale, individuals are asked how safe they feel during these activities and they are asked to give a score between 1 and 10 (1 = safest, 10 = least safe). When all scores are added in scale, a total score between 0-100 is obtained. High scores indicate that the individual's fear of falling increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)